CLINICAL TRIAL: NCT04288167
Title: Biochemical Diagnostics of Mild Traumatic Brain Injury (TBI) and Concussion in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medicortex Finland Oy (Industry)
Collaborators: Satasairaala (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: T257/2019
Record Dates: First submitted 2020-02-13; First posted 2020-02-28 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Specimen Handling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The laboratories will analyze the samples blinded, without knowing whether the sample was from an injured patient or a healthy control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with suspected brain injury (Experimental): This arm will consist of up to 30 pediatric patients who entered the Emergency Room and who are suspected of having mild traumatic brain injury. Two sample sets will be collected within the first 10 hours from the injury.
  Interventions: Diagnostic Test: Sample collection
- Healthy controls (Active Comparator): This arm will consist of up to 30 healthy control subjects, the samples of whom will be compared to the samples of brain injury patients (Arm 1). One sample set will be collected from healthy children without any known brain injury.
  Interventions: Diagnostic Test: Sample collection

INTERVENTIONS:
Diagnostic Test: Sample collection — Samples of urine and saliva will be collected from participants using customary sample collection means.

SUMMARY:
The study will enroll children and adolescents (0 - 17 years) suspected of having concussion or mild traumatic brain injury (TBI). Samples of urine and saliva will be collected from the patients as well as from corresponding age- and gender-adjusted healthy controls.

DETAILED DESCRIPTION:
The collected samples will be alienated to the Sponsor who will perform biochemical studies to identify and measure from the samples relative level of the brain injury-specific biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* The subject is suspected of having an isolated mild TBI (Glasgow Coma Score 13 - 15)
* No more that 6 hours elapsed from the incident of injury at the first sampling
* The patient is conscious
* Informed consent received from the legal guardian, and the subject him-/herself when literate and capable of understanding study measures

Exclusion Criteria:

* More than 6 hours elapsed from the injury, or unknown time of trauma
* Multi-trauma patient
* History of head injury, seizures or stroke within three preceding months
* Chronic neurodegenerative, metabolic or autoimmune disease
* Known existing neurological condition

Ages: 1 Minute to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Biomarker levels | 12 months
  Quantitative measurement of the novel glycan-based biomarker using a lectin-binding assay
Biomarker profiles | 12 months
  Characterization of different glycan structures present in the sample by mass spectrometry analysis

CONTACTS AND LOCATIONS:
Overall Officials: Sari Malmi, MD, Principal Investigator — Satasairaala
Locations (1):
- Satakunta Central Hospital, Pori, Finland

IPD SHARING:
Plan to Share IPD: No
Individual participant data shall not be shared to outside of the study.